CLINICAL TRIAL: NCT02167087
Title: Sentinel Node Mapping With Indocyanine Green in Colon Cancer: a Feasibility Trial and a Descriptive Serie.
Acronym: SENSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ismail Gögenür (Other)
Responsible Party: Sponsor-Investigator, Ismail Gögenür, Professor, DMSc, MD, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SENSE2014
Record Dates: First submitted 2014-06-06; First posted 2014-06-18 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Colon Cancer; Lymphatic Metastasis
Keywords: Sentinel node mapping; lymphatic mapping; lymphatic metastasis; Aberrant lymphatic drainage; indocyanine green; ICG; near infrared; colon cancer; laparoscopic surgery
MeSH Terms: conditions — Colonic Neoplasms; Lymphatic Metastasis | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sentinel node mapping (Experimental): Sentinel node mapping with indocyanine green injected orally and anally to the tumor.
  Interventions: Procedure: Sentinel node mapping

INTERVENTIONS:
Procedure: Sentinel node mapping — Through transabdominal access via laparoscopic ports indocyanine green solution is injected around the tumor (25 mg indocyanine green dissolved in 9 ml sterile water and 1 ml 20% human albumin). This is done by the construction of two small boluses of 0.5 mL each into the colonic wall just orally and anally to the tumor margin, but not within the tumor itself. When the bolus is injected the fluorescence is controlled and after 20 minutes the surgeon looks for sentinel nodes in a standardized manner.
  Other Names: Karl Storz ICG system, to visualize the fluorescence; Indocyanine green, PULSION medical systems.; Single use aspiration needle, NA-220H-8025 from Olympus.

SUMMARY:
This study is a clinical feasibility trial that will contribute to the clarification of whether sentinel node mapping with indocyanine green (ICG) provides a better basis for staging of colorectal cancer.

DETAILED DESCRIPTION:
The patients assigned for colon cancer will be operated as planned using laparoscopic techniques and the operation follows the normal procedure, in addition a sentinel node mapping is performed.

Indocyanine green is injected around the tumor by laparoscopic technique, the fluorescence is controlled and after 20 minutes the surgeon looks for sentinel nodes in a standardized manner. In the meantime, the surgeon proceeds with the operation as usual, except that the mesocolon can be resected only after sentinel node mapping has been performed.

After surgery the surgeon and the pathologist inspect the resected colon together and agree on D1, D2 and D3 margins. Any marked sentinel node(s) is verified and the location is checked on the colon diagram on the case report form. In addition, an ex vivo sentinel node mapping will be performed by the pathologist right after the surgery has ended. This is done to investigate if it is the same lymph nodes there will be identified by ex vivo as by intraoperative (in vivo) sentinel node mapping.

The lymph nodes in the resected colon and mesocolon are all analysed. Sentinel nodes and an equal number of randomly chosen non-sentinel nodes will be analysed further with additional sections and immune histochemistry.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients above 18 years of age scheduled for laparoscopic colon cancer surgery in the department of Surgery, Herlev Hospital or Roskilde Hospital.

Exclusion Criteria:

* iodine allergy
* Poor kidney function (as it imply an increased risk of allergic reaction), estimated glomerular filtration rate should be above 40 ml/min.
* Liver cirrhosis, Child-Pugh-score B and C [14]
* Pregnancy and lactation
* Previous anaphylactic reaction to a dye injection
* Previous abdominal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Number of procedures with successful identification of sentinel nodes | day 1
  Sentinel nodes is defined as the lymph node, first in line, draining from the cancer.

SECONDARY OUTCOMES:
Number of sentinel nodes identified during surgery and their localization | day 1
Number of sentinel nodes identified by ex vivo sentinel node mapping | week 1
Malignant status of the sentinel node(s) | week 1
Malignant status of the lymph nodes | week 1
Number of cases with negative sentinel node, but positive non-sentinel node | week 1
Localization of sentinel nodes with metastasis | week 1
Localization of lymph nodes with metastasis according to D1, D2 and D3 resection lines and if they are within 1 cm from a sentinel node | week 1
Number of cases where the sentinel node procedure has changed the clinical course of the patient | week 1
  if staging and oncological treatment are changed because of the procedure
Number of procedures where the procedure is stopped due to technical reasons | day 1
Registration of possible side effects occurring due to the use of indocyanine green | day 1
Number of sentinel nodes identified by only one of the sentinel node mapping techniques | week 1
Total number of lymph nodes | week 1
Localization of the identified sentinel nodes, and whether or not they are included within the normal resection lines | week 1

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Gögenur, Professor, Principal Investigator — Professor at University Hospital Køge
Locations (1):
- Herlev Hospital, Herlev, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: Undecided